CLINICAL TRIAL: NCT05552014
Title: Research on the Efficacy Mechanism of Natural Psychotherapy for Neurosis
Brief Title: Study on the Efficacy Mechanism of Natural Psychotherapy for Neurosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Professor, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASPsy5
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive-compulsive disorder; natural psychotherapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient was assigned to either the intervention group or the control group, but the control group would also receive treatment after a two-month waiting period. Therefore, the patient was only informed whether they would be participating in the first or second intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Natural Psychotherapy (Active Comparator): Intervention using natural psychotherapy for OCD patients for two to three hours once a week for eight weeks
  Interventions: Behavioral: Natural Psychotherapy
- Mental Health Education (Placebo Comparator): Mental health education was given to another group of OCD patients for two hours once a week for eight weeks
  Interventions: Behavioral: Mental Health Education

INTERVENTIONS:
Behavioral: Natural Psychotherapy — Natural psychotherapy is based on "Morita therapy" and is a psychotherapy that fully reflects the characteristics of Chinese culture, taking into account the Chinese cultural background and actual clinical characteristics.
  Arms: Natural Psychotherapy
Behavioral: Mental Health Education — Mental Health Education Seminar
  Arms: Mental Health Education

SUMMARY:
explore objective indicators of the efficacy of natural psychotherapy in the treatment of disorders such as obsessive-compulsive disorder

DETAILED DESCRIPTION:
1. To evaluate the cognitive function, Cognitive control, emotion and other aspects of neurosis patients, and to understand and master the cognitive behavior indicators of this population.
2. Investigate the pathological mechanism of neurotic patients from the aspects of EEG/fMRI and biology.
3. To investigate the therapeutic effect of natural psychotherapy on cognitive impairment and related mood, sleep and symptom intervention in neurotic patients. In order to achieve the symptoms of neurosis patients, cognitive impairment and related mood and sleep intervention and promotion, while providing a scientific basis for neurosis rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* were between 16 and 55 years old;
* were diagnosed with OCD by an experienced psychiatrist utilizing the Structured Clinical Interview for DSM-5 (SCID);
* had an illness duration of at least 12 months;
* were able to participate in the entire trial and face-to-face on-site assessment

Exclusion Criteria:

* pregnant or breastfeeding;
* suffered from organic brain diseases or severe physical illness;
* had a history of substance or alcohol abuse
* were at high risk of suicide

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Obsessive-compulsive symptoms | Baseline, week 4, week 8
  Using the score of Yale-Brown Obsessive-Compulsive Scale as the primary outcome, a decrease in score of ≥35% was considered a 'response to treatment', also referred to as a 'full response', and a decrease in score of ≥25% was considered a 'partial response'

SECONDARY OUTCOMES:
Self-reported obsessive-compulsive symptoms | Baseline, week 4, week 8
  The reduction rate of the score of Obsessive-Compulsive Inventory-Revised (OCI-R), a self-rating scale of OCD symptoms severity, was employed as a secondary outcome
Cognitive inhibition | Baseline, week 8
  Cognitive inhibition was assessed using the emotional color-word Stroop task. The emotional Stroop task is a type of being Widely used cognitive inhibition assessment tools. The longer the reaction time, the worse the cognitive inhibition ability.
Behavioral inhibition | Baseline, week 8
  Behavioral inhibition was assessed using the emotional stop signal task (SST). The emotional SST task is a type of being Widely used behavioral inhibition assessment tools. Among them, the greater the SSRT, the worse the behavioral inhibition ability.
ERP components associated with cognitive function | Baseline, week 8
  To explore the ERP component analysis related to cognitive inhibition and Behavioral inhibition in obsessive-compulsive disorder (OCD) by event related potential (ERP) analysis
rest fMRI in Obsessive-compulsive patients | Baseline, week 8
  The changes of resting-state functional connectivity were analyzed in patients with OCD before and after intervention. Resting-state functional connectivity：FC(Functional connectivity). Resting-state functional brain imaging data were collected using a GE 3.0T magnetic resonance scanner (GE Discovery MR750) at the Brain Imaging Center, Institute of Psychology, Chinese Academy of Sciences.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Y Zhang, M.D, Ph.D, Principal Investigator — Institute of Psychology, Chinese Academy of Science
Locations (2):
- China (2):
  - Anhui Mental Health Center, Hefei, Anhui
  - Institute of Psychology, Chinese Academy of Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Data with be available on request